CLINICAL TRIAL: NCT05989009
Title: Essential Long-chain Polyunsaturated Fatty Acids Quantitation in Breast Milk Samples At Different Gestational Ages
Brief Title: Analysis of Lipids in Human Milk At Different Gestational Ages
Status: Completed | Type: Observational
Sponsor: Ospedale Buon Consiglio Fatebenefratelli (Other)
Collaborators: University of Salerno (Other)
Responsible Party: Principal Investigator, Giuseppe De Bernardo, Head of Department of Woman and Child, Ospedale Buon Consiglio Fatebenefratelli
Other Study IDs: 1669/CE Lazio 1
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-08

CONDITIONS: Breast Milk Collection
Keywords: newborn; breast milk; fatty acid; gestational age
MeSH Terms: conditions — Breast Milk Expression | interventions — Lactation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Women < 32 weeks of gestational age: Women that delivered before 32 weeks of gestational age
  Interventions: Other: Breastfeeding
- Women between 32 and 36,6 weeks of gestational age: Women that delivered between 32 and 36,6 weeks of gestational age
  Interventions: Other: Breastfeeding
- Women > 37 weeks of gestational age: Women that delivered after 37 weeks of gestational age
  Interventions: Other: Breastfeeding

INTERVENTIONS:
Other: Breastfeeding — Mothers will breastfeed their newborns

SUMMARY:
Various studies have shown that the milk of a preterm infant differs from that of a term infant in the composition of micronutrients, vitamins, macronutrients, carbohydrates and proteins. The study of lipidomic is of particular interest because the role of fatty acids is known both as essential constituents of cell membranes and as molecules actively involved in energy metabolism. The study of human milk would offer the advantage of offering the best type of nutrition for the newborn at each specific period of life, in the event of a lack of mother's milk.

DETAILED DESCRIPTION:
Mother's milk is the best food for the newborn as it is the only one capable of providing species-specific nutrition, guaranteeing everything necessary for the growth and maturation of a child. Mother's milk has the property of satisfying metabolic needs by changes in the composition of nutrients, which are different at each stage of life. Various studies have shown that the milk of a preterm infant differs from that of a term infant in the composition of micronutrients, such as vitamins, macronutrients, carbohydrates and proteins. The metabolomic study of human milk would offer the advantage of offering the best type of nutrition for the newborn at each specific period of life, in the event of a lack of mother's milk. This is particularly important in a Neonatal Intensive Care Unit, where it is essential to ensure timely adequate enteral nutrition. This is possible if a bank of donated human milk is available. The study of lipidomics is of particular interest, as the role of fatty acids is known both as essential constituents of cell membranes and as molecules actively involved in energy metabolism. Therefore, the benefit deriving from an adequate dietary intake in a constantly evolving organism such as that of a newborn is extremely important.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have given birth in hospital at any gestational age
* Written informed consent
* BMI 18.50-24.99 Kg/m2
* Varied and balanced maternal diet without restrictions
* Weight gain during pregnancy up to 12kg

Exclusion Criteria:

* Food intolerance
* Celiac disease
* Vegan or vegetarian diet
* Diet with the exclusion of milk and derivatives
* Diagnosis of metabolic diseases
* Taking medicines during pregnancy
* Withdrawal of informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: They were enrolled mothers that delivered at Buon Consiglio Fatebenefratelli Hospital, Napoli
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 7 days after delivery
  To assess the concentrations of α-Linoleic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 7 days after delivery
  To assess the concentrations of Eicosapentaenoic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 7 days after delivery
  To assess the concentrations of Docosahexaenoic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 7 days after delivery
  To assess the concentrations of Arachidonic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 7 days after delivery
  To assess the concentrations of Linoleic acid (µg/mL) in human milk

SECONDARY OUTCOMES:
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 1 month after delivery
  To assess the concentrations of α-Linoleic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 1 month after delivery
  To assess the concentrations of Eicosapentaenoic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 1 month after delivery
  To assess the concentrations of Docosahexaenoic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 1 month after delivery
  To assess the concentrations of Arachidonic acid (µg/mL) in human milk
Quantification of essential long-chain polyunsaturated fatty acids in human milk | 1 month after delivery
  To assess the concentrations of Linoleic acid (µg/mL) in human milk

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Bernardo, MD, Principal Investigator — Ospedale Buon Consiglio Fatebenefratelli
Locations (2):
- Italy (2):
  - Department of Pharmacy, University of Salerno, Salerno, Naples
  - Department of Woman and Child, Buon Consiglio Fatebenefratelli Hospital, Napoli, Napoli